CLINICAL TRIAL: NCT03387605
Title: Effect of Ivabradine on Heart Rate and Hemodynamics in Patients With Stage D Heart Failure (HF)/Cardiogenic Shock on Dobutamine Treatment
Brief Title: Effect of Ivabradine in Stage D HF/Cardiogenic Shock Patients on Dobutamine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Eugenia Raichlin, Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 209939
Record Dates: First submitted 2017-12-15; First posted 2018-01-02 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure; Cardiogenic Shock; Tachycardia
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic; Tachycardia | interventions — Ivabradine

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blind, Placebo Controlled single center study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivabradine (Active Comparator): Initiation at dose 5 mg PO x 1 dose and further increased in 12 hours to 7.5 mg PO twice per day if patient is stable with mean BP≥ 60 mmHg, systolic blood pressure ≥ 90 mmHg and HR ≥100 bpm
  Interventions: Drug: Ivabradine
- Placebo (Placebo Comparator): Matching placebo given PO twice per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — ivabradine or placebo given orally 2 times daily for 72 hours
  Other Names: Corlanor
  Arms: Ivabradine
Drug: Placebo — matching placebo given 2 times daily for 72 hours
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, single center trial to study of the effects of Ivabradine vs. Placebo on patients hospitalized for Stage D heart failure (HF)/ and cardiogenic shock (CS) who will require continuous infusion of Dobutamine and have developed sinus tachycardia (ST) (heart rate >100 beats/min).

The aim of the study will be to assess the potential of Ivabradine to slow ST and improve hemodynamics in patients with stage D HF/CS on Dobutamine treatment.

DETAILED DESCRIPTION:
This study will explore the hypothesis that Ivabradine will decrease heart rate (HR) and improve hemodynamics in patients with advanced HF on inotropic treatment. This is a randomized, double blind, single center trial will include 40 consecutive patients admitted for Stage D HF/ CS who will require continuous infusion of Dobutamine and will develop ST (HR >100 beats/min).

Eligible patients will be randomized (1:1) using blocked randomization with random block sizes of 2 or 4 to start Ivabradine versus placebo. The procedure of randomization to receive either Ivabradine or placebo twice daily will be performed by computerized sequence generation. The hospital pharmacies will be responsible for drug randomization and dispensing, and the investigators and the patients will be blinded to the treatment option.

Ivabradine will be started 3 hours after Dobutamine initiation at dose 5 mg and further increased in 12 hours to 7.5 mg bid if patient is stable with mean BP≥ 60 mmHg, systolic blood pressure ≥ 90 mmHg and HR ≥100 bpm. Increase of Ivabradine dosage will be individually stopped for reasons of safety if three episodes of minimal HRs of less than 70 beats per minute, or a drop in mean blood pressure < 60 mmHg or systolic blood pressure < 80 mmHg occur.

HR, blood pressure and invasive hemodynamics will be monitored, along with standard right heart cath and echocardiogram measurements obtained.

Patients will be followed for a total of 72 hours. The adverse events that will be collected include bradycardia, defined as a heart rate less than 70 bpm, hypotension defined as a systolic blood pressure less than 80 mmHg and any side effect requiring drug discontinuation or dose adjustment. Review of laboratory including renal, hepatic and hematologic counts will be reviewed for any significant changes due to the use of Ivabradine.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent for the study
* Have current diagnosis of Ischemic and/or non-ischemic cardiomyopathy
* Left ventricular ejection fraction (LVEF) < 30% by echo during the screening
* Sinus rhythm with HR ≥100 bpm
* Systolic blood pressure ≥ 90 mmHg assessed by cuff sphygmomanometer
* CI < 2.2 L/min/m2
* Current symptom(s) of HF (New York Heart Association (NYHA) class IV) at Screening.
* Absence of hypovolemia, defined as a central venous pressure ≥10 mmHg and pulmonary capillary occlusion pressure ≥15 mmHg before administration of Dobutamine

Exclusion Criteria:

* Respiratory support with mechanical ventilation
* Circulatory mechanical support
* Atrial pacing with the presence of sick sinus syndrome or sino-atrial block
* Second or third degree atrioventricular (AV) block,
* Atrial fibrillation/flutter
* Amiodarone treatment
* Ventricular tachycardia
* Acute coronary syndrome
* Bilirubin > 2.5
* Alanine aminotransferase (ALT) >60 IE/L,
* Serum creatinine >2.5 g/ml)
* Fever and significant infection
* Pregnancy
* Anemia, Hgb < 9.0
* Patients required treated with severe cytochrome CYP3A4 inhibitors drugs Concomitant use of strong CYP3A4 inhibitors will be avoided during the study period

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Heart rate | 72 hours
  Heart rate will be measured and any changes noted

SECONDARY OUTCOMES:
cardiac index | 72 hours
  cardiac index will be assessed by pulmonary artery catheter and any changes noted
plasma brain natriuretic peptide (BNP) level | 72 hours
  Labs will be drawn for plasma BNP blood test and any changes noted

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Raichlin, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reynolds HR, Hochman JS. Cardiogenic shock: current concepts and improving outcomes. Circulation. 2008 Feb 5;117(5):686-97. doi: 10.1161/CIRCULATIONAHA.106.613596. No abstract available. PMID 18250279
- [Background] Vasquez A, Kern KB, Hilwig RW, Heidenreich J, Berg RA, Ewy GA. Optimal dosing of dobutamine for treating post-resuscitation left ventricular dysfunction. Resuscitation. 2004 May;61(2):199-207. doi: 10.1016/j.resuscitation.2004.01.002. PMID 15135197
- [Background] Leier CV, Webel J, Bush CA. The cardiovascular effects of the continuous infusion of dobutamine in patients with severe cardiac failure. Circulation. 1977 Sep;56(3):468-72. doi: 10.1161/01.cir.56.3.468. PMID 884803
- [Background] Metra M, Nodari S, D'Aloia A, Muneretto C, Robertson AD, Bristow MR, Dei Cas L. Beta-blocker therapy influences the hemodynamic response to inotropic agents in patients with heart failure: a randomized comparison of dobutamine and enoximone before and after chronic treatment with metoprolol or carvedilol. J Am Coll Cardiol. 2002 Oct 2;40(7):1248-58. doi: 10.1016/s0735-1097(02)02134-4. PMID 12383572
- [Background] Wynsen JC, O'Brien PD, Warltier DC. Zatebradine, a specific bradycardic agent, enhances the positive inotropic actions of dobutamine in ischemic myocardium. J Am Coll Cardiol. 1994 Jan;23(1):233-41. doi: 10.1016/0735-1097(94)90526-6. PMID 8277087
- [Background] Aidonidis I, Brachmann J, Rizos I, Zacharoulis A, Stavridis I, Toutouzas P, Kubler W. Electropharmacology of the bradycardic agents alinidine and zatebradine (UL-FS 49) in a conscious canine ventricular arrhythmia model of permanent coronary artery occlusion. Cardiovasc Drugs Ther. 1995 Aug;9(4):555-63. doi: 10.1007/BF00878087. PMID 8547205
- [Background] Hettrick DA, Pagel PS, Lowe D, Tessmer JP, Warltier DC. Increases in inotropic state without change in heart rate: combined use of dobutamine and zatebradine in conscious dogs. Eur J Pharmacol. 1996 Dec 5;316(2-3):237-44. doi: 10.1016/s0014-2999(96)00688-7. PMID 8982692
- [Background] Neustein SM, Dimich I, Shiang H, Mezrow C. Role of zatebradine and propranolol in attenuation of tachycardia produced by dobutamine in pigs. Acta Anaesthesiol Scand. 1997 Aug;41(7):849-52. doi: 10.1111/j.1399-6576.1997.tb04799.x. PMID 9265927
- [Background] Zhang Y, Mazgalev TN. Cardiac vagal stimulation eliminates detrimental tachycardia effects of dobutamine used for inotropic support. Ann Thorac Surg. 2009 Jul;88(1):117-22. doi: 10.1016/j.athoracsur.2009.04.009. PMID 19559207
- [Background] DiFrancesco D, Camm JA. Heart rate lowering by specific and selective I(f) current inhibition with ivabradine: a new therapeutic perspective in cardiovascular disease. Drugs. 2004;64(16):1757-65. doi: 10.2165/00003495-200464160-00003. PMID 15301560
- [Background] Fox K, Ford I, Steg PG, Tendera M, Ferrari R; BEAUTIFUL Investigators. Ivabradine for patients with stable coronary artery disease and left-ventricular systolic dysfunction (BEAUTIFUL): a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Sep 6;372(9641):807-16. doi: 10.1016/S0140-6736(08)61170-8. Epub 2008 Aug 29. PMID 18757088
- [Background] Swedberg K, Komajda M, Bohm M, Borer JS, Ford I, Dubost-Brama A, Lerebours G, Tavazzi L; SHIFT Investigators. Ivabradine and outcomes in chronic heart failure (SHIFT): a randomised placebo-controlled study. Lancet. 2010 Sep 11;376(9744):875-85. doi: 10.1016/S0140-6736(10)61198-1. PMID 20801500
- [Background] Henri C, O'Meara E, De Denus S, Elzir L, Tardif JC. Ivabradine for the treatment of chronic heart failure. Expert Rev Cardiovasc Ther. 2016;14(5):553-61. doi: 10.1586/14779072.2016.1165092. Epub 2016 Mar 28. PMID 26967048
- [Background] Tardif JC, O'Meara E, Komajda M, Bohm M, Borer JS, Ford I, Tavazzi L, Swedberg K; SHIFT Investigators. Effects of selective heart rate reduction with ivabradine on left ventricular remodelling and function: results from the SHIFT echocardiography substudy. Eur Heart J. 2011 Oct;32(20):2507-15. doi: 10.1093/eurheartj/ehr311. Epub 2011 Aug 29. PMID 21875858
- [Background] Fang Y, Debunne M, Vercauteren M, Brakenhielm E, Richard V, Lallemand F, Henry JP, Mulder P, Thuillez C. Heart rate reduction induced by the if current inhibitor ivabradine improves diastolic function and attenuates cardiac tissue hypoxia. J Cardiovasc Pharmacol. 2012 Mar;59(3):260-7. doi: 10.1097/FJC.0b013e31823e5e01. PMID 22075752
- [Background] Mulder P, Barbier S, Chagraoui A, Richard V, Henry JP, Lallemand F, Renet S, Lerebours G, Mahlberg-Gaudin F, Thuillez C. Long-term heart rate reduction induced by the selective I(f) current inhibitor ivabradine improves left ventricular function and intrinsic myocardial structure in congestive heart failure. Circulation. 2004 Apr 6;109(13):1674-9. doi: 10.1161/01.CIR.0000118464.48959.1C. Epub 2004 Feb 23. PMID 14981003
- [Background] Boldt A, Gergs U, Ponicke K, Simm A, Silber RE, Neumann J. Inotropic effects of ivabradine in the mammalian heart. Pharmacology. 2010;86(5-6):249-58. doi: 10.1159/000320454. Epub 2010 Oct 21. PMID 20962545
- [Background] Reil JC, Tardif JC, Ford I, Lloyd SM, O'Meara E, Komajda M, Borer JS, Tavazzi L, Swedberg K, Bohm M. Selective heart rate reduction with ivabradine unloads the left ventricle in heart failure patients. J Am Coll Cardiol. 2013 Nov 19;62(21):1977-1985. doi: 10.1016/j.jacc.2013.07.027. Epub 2013 Aug 7. PMID 23933545
- [Background] De Ferrari GM, Mazzuero A, Agnesina L, Bertoletti A, Lettino M, Campana C, Schwartz PJ, Tavazzi L. Favourable effects of heart rate reduction with intravenous administration of ivabradine in patients with advanced heart failure. Eur J Heart Fail. 2008 Jun;10(6):550-5. doi: 10.1016/j.ejheart.2008.04.005. Epub 2008 May 16. PMID 18486549
- [Background] Cavusoglu Y, Mert U, Nadir A, Mutlu F, Morrad B, Ulus T. Ivabradine treatment prevents dobutamine-induced increase in heart rate in patients with acute decompensated heart failure. J Cardiovasc Med (Hagerstown). 2015 Sep;16(9):603-9. doi: 10.2459/JCM.0000000000000033. PMID 24922198
- [Background] Roubille F, Lattuca B, Busseuil D, Leclercq F, Davy JM, Rheaume E, Tardif JC. Is ivabradine suitable to control undesirable tachycardia induced by dobutamine in cardiogenic shock treatment? Med Hypotheses. 2013 Aug;81(2):202-6. doi: 10.1016/j.mehy.2013.05.002. Epub 2013 May 26. PMID 23719030
- [Background] Franke J, Schmahl D, Lehrke S, Pribe R, Bekeredjian R, Doesch AO, Ehlermann P, Schnabel P, Katus HA, Zugck C. Adjuvant Use of Ivabradine in Acute Heart Failure due to Myocarditis. Case Rep Med. 2011;2011:203690. doi: 10.1155/2011/203690. Epub 2011 Sep 27. PMID 21966292
- [Background] Link A, Reil JC, Selejan S, Bohm M. Effect of ivabradine in dobutamine induced sinus tachycardia in a case of acute heart failure. Clin Res Cardiol. 2009 Aug;98(8):513-5. doi: 10.1007/s00392-009-0038-9. Epub 2009 Jun 23. No abstract available. PMID 19547907
- [Background] Vitale D, De Santis V, Guarracino F, Fontana A, Pellegrini F, Tritapepe L. Use of ivabradine in catecholamine-induced tachycardia after high-risk cardiac surgery. Clin Res Cardiol. 2010 Dec;99(12):853-5. doi: 10.1007/s00392-010-0208-9. Epub 2010 Sep 7. No abstract available. PMID 20821020
- [Background] Gallet R, Ternacle J, Damy T, Guendouz S, Bremont C, Seemann A, Gueret P, Dubois-Rande JL, Lim P. Hemodynamic effects of Ivabradine in addition to dobutamine in patients with severe systolic dysfunction. Int J Cardiol. 2014 Sep 20;176(2):450-5. doi: 10.1016/j.ijcard.2014.07.093. Epub 2014 Aug 1. PMID 25129291
- [Background] Borlaug BA, Nishimura RA, Sorajja P, Lam CS, Redfield MM. Exercise hemodynamics enhance diagnosis of early heart failure with preserved ejection fraction. Circ Heart Fail. 2010 Sep;3(5):588-95. doi: 10.1161/CIRCHEARTFAILURE.109.930701. Epub 2010 Jun 11. PMID 20543134
- [Background] Borlaug BA, Kass DA. Ventricular-vascular interaction in heart failure. Heart Fail Clin. 2008 Jan;4(1):23-36. doi: 10.1016/j.hfc.2007.10.001. PMID 18313622
- See also: article: Safety, tolerability and efficacy of ivabradine for control of sinus tachycardia in patients undergoing inotropic therapy — http://medicontenidosporcile.files.wordpress.com/2016/03/curr-reserch-cardiol.pdf